CLINICAL TRIAL: NCT01772407
Title: Right Colon Cancer: Laparoscopic Surgery Versus Open Surgery, Costs, Mortality, Morbidity and Quality of Life
Brief Title: Laparoscopic Surgery Equivalent to Open Surgery in Right Colon Cancer Surgery?
Acronym: CHIRCOL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: STIC ICO711
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2016-05

CONDITIONS: Colon Cancer
Keywords: Colon Cancer Surgery; Laparoscopy; Open surgery; Costs; Mortality; Morbidity; Quality of life
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: laparoscopic surgery in right colon cancer operations
- 2: open surgery in right colon cancer operations

SUMMARY:
The primary goal of this study is to compare in the long-term costs of laparoscopic or open right colectomy in patients sustaining a colon cancer controling for the carcinologic equivalence of the two surgical strategies. The secondary goals to compare long-term mortality, morbidity as well as quality of life of the two groups.The present study is an prospective multicentric observational trial taking into account the usual surgical strategy of every centers

DETAILED DESCRIPTION:
The aim of the present study is to compare in the long-term costs of laparoscopic and open right cancer colectomy as well as the mortality the morbidity and the quality of life of the operated patients.

The number of patients need to get a 54% power is 300. The average number of patients/surgical center is approximately 27 in 14 surgical centers.

The proposed undertaking of every patient is fully identical to that which is usually proposed by the surgical center in charge of the patient (i.d. 7 centers will perform laparoscopic procedures and 7 centers open procedure according to their usual practice).

A complete information leaflet will be given to the patients during the first consultation which will correspond to the enrollment day.

The preoperative, intraoperative and postoperative period will be in complete accordance with the usual care of the center.

The baseline demographics and conditions as well as the perioperative items and the postoperative occurrences will be recorded through a prior designed e-questionnaire.

The follow-up encompass 5 postoperative consultations:1 month, 6 ,12 ,18 and 24 months.

On every consultation the patient will fill a very simple validated quality of life questionnaire (EORTC,QLQ.C30) an give back a weekly journal reporting the potentially arising medical and surgical events.

Globally the comparative analysis of the costs ,the mortality ,the morbidity, the quality of life ot the patients undergoing either a laparoscopic or a open right colectomy for cancer will be performed controling for the carcinologic equivalence of the two surgical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old <= 80 years old
* Right colon cancer < T4 without metastasis
* <T4 N0M0

Exclusion Criteria:

* Pregnant patient
* T4 cancer
* Metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Right colon cancer < T4 without metastasis needing colectomy
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cost during the 2 postoperative years | during the 2 postoperative years

SECONDARY OUTCOMES:
Mortality, morbidity and quality of life during the 2 postoperative years | during the 2 postoperative years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Hannoun, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié-Salpetrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No